CLINICAL TRIAL: NCT05835570
Title: A Single-arm, Open-label, Single-center Clinical Study to the Evaluation of Integrin αvβ6-targeted Positron Emission Tomography (PET) for Malignant Tumors
Brief Title: Integrin αvβ6-targeted PET in Malignant Tumors
Status: Recruiting | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Yong He, Chief of Department of Nuclear Medicine, Zhongnan Hospital
Other Study IDs: ZNYYHYXK0003
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Malignant Neoplasm; PET/CT; Non-Small Cell Lung Cancer; Breast Cancer, Metastatic
Keywords: Non-small cell lung cancer; Breast cancer; Integrin-αvβ6; [68Ga]Ga-Trivehexin; Malignant tumors
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Neoplasm Metastasis | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Integrin αvβ6-targeted PET in malignant tumors: Participants: newly diagnosed malignant tumor confirmed by pathology or suspected lung cancer. Interventions: Participant who conforms to the inclusion criteria will undergo 18F-FDG and 68Ga-Trivehexin PET/CT scans within 1 week.
  Interventions: Participant who conforms to the inclusion criteria will undergo 18F-FDG and 68Ga-Trivehexin PET/CT scans within 1 week.
  Objectives: This study aims to assess and compare the diagnostic performance of 68Ga-Trivehexin and 18F-FDG PET/CT for the detection of primary tumors, mediastinal lymph nodes and distant metastases, and to explore the correlation between 68Ga-Trivehexin accumulation and immunohistochemical β6 expression in NSCLC.
  Interventions: Diagnostic Test: PET/CT scans

INTERVENTIONS:
Diagnostic Test: PET/CT scans — Diagnostic Test: For 68Ga-Trivehexin PET/CT, no special preparation was required. Approximately 50 min after an i.v. administration of [68Ga]Ga-Trivehexin with a dose of 1.85-2.22 MBq/kg, and the PET acquisition time was 2.5 min per bed.

SUMMARY:
Malignant tumors are a significant health threat with high incidence and mortality rates, and molecular imaging is crucial for early diagnosis, staging, prognosis evaluation, and therapeutic efficacy assessment. 18F-FDG PET imaging is widely used, but has limitations. Integrin αvβ6 is a promising target for tumor-targeted imaging, as it is only expressed in cancerous or reconstructed epithelial cells. A new PET probe, 68Ga-Trivehexin, targeting integrin αvβ6 has been developed with better affinity and selectivity than previous probes. Clinical data supports its safety and metabolic stability, and future research will explore its diagnostic and staging value in different types of tumors, providing a new and precise evaluation method for malignant tumors.

DETAILED DESCRIPTION:
Malignant tumors are a significant disease that threatens human health and life, with high incidence and mortality rates. Molecular imaging plays an important role in the early diagnosis, staging, prognosis evaluation, and therapeutic efficacy assessment of major diseases such as tumors. Currently, 18F-FDG PET imaging is the most widely used molecular imaging, but there are still problems such as physiological uptake, false negatives, and false positives. It is urgent to explore and develop a new type of tumor-targeting PET imaging.

Integrins are key members of the cell adhesion molecular family and play a central role in regulating cell-cell and cell-extracellular matrix interactions. They are highly expressed in a variety of malignant tumors and plays a vital role in the angiogenesis, invasion and metastasis of tumors, and the regulation of immune microenvironment. As such, integrins have emerged as potential targets for tumor-specific imaging. To date, PET tracers targeting integrin αvβ3 have been extensively studied for imaging tumor neovascularization. However, this integrin subtype also shows certain expression in normal tissue endothelial cells, posing a challenge to its clinical value as a specific marker for tumor imaging. In contrast, integrin αvβ6, another subtype of integrin known as "cancer integrin", is specifically expressed in epithelial-derived tumor cells, whereas it hardly expressed in human healthy tissues. Therefore, integrin αvβ6 has gained attention as an attractive and promising biomarker.

In the past decade, some integrin αvβ6-targeting PET tracers have been synthesized, but these agents have shown relatively low affinity and specificity, with high nonspecific uptake in the gastrointestinal tract, which hinders their clinical translation. Recently, Quigley et al. introduced a novel αvβ6-targeted trimeric probe based on a cyclic peptide c[YRGDLAYp(NMe)K], named 68Ga-Trivehexin. This probe demonstrated favorable characteristics, including excellent targeting affinity (IC50 = 0.047 nM), enhanced tumor uptake, and longer retention time in preclinical study. The preliminary results from PET imaging in 4 cancer patients further demonstrated intense 68Ga-Trivehexin accumulation in head and neck squamous cell carcinoma, parotid adenocarcinoma and pancreatic ductal adenocarcinoma; moreover, there was almost no physiological uptake in normal tissues and organs, such as stomach, intestine, liver, and lung, except for kidney (the excretory organ), resulting in an excellent tumor-to-background ratio.

The safety and metabolic stability of 68Ga-Trivehexin targeting integrin αvβ6 are currently supported by clinical data, and this project will further expand its application in various malignant tumors, clarify its diagnostic and staging value in different types of tumors, and qualitative and quantitative characteristics. This project is expected to provide a new and precise evaluation method for malignant tumors to compensate for the shortcomings of current imaging methods.

ELIGIBILITY:
Inclusion Criteria:

* Participants with newly diagnosed malignant tumor confirmed by pathology or suspected lung cancer;
* Age ≥18 years, regardless of gender;
* No prior anti-tumor therapy (e.g., chemotherapy, radiotherapy, targeted therapy, or immunotherapy) before PET/CT;
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-1;
* Female subjects of reproductive age, male subjects and their partners agree to use reliable contraceptive measures (e.g., abstinence, birth control pills, injectable contraceptives, or subcutaneous contraceptive implants) until 6 months after the completion of the study;
* Participants should voluntarily consent to the clinical trial, and have the ability to understand and sign an informed consent form.

Exclusion Criteria:

* Known allergy to injection or its excipients;
* Severe liver or renal dysfunction;
* Claustrophobia or other psychiatric disorders;
* History of other malignant tumors;
* Participation in another clinical trial within 30 days prior to PET/CT scan;
* Pregnant or breastfeeding women;
* Refusal to participate or request for withdrawing from the clinical study;
* Other conditions deemed unsuitable for inclusion by investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in-patinets
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The diagnostic sensitivity and specificity of 68Ga-Integrin αvβ6 PET/CT in the staging of malignant tumors | 2 years
  The diagnostic performance of [68Ga]Ga-Trivehexin PET/CT and [18F]-FDG PET/CT for initial staging will be evaluated and compared using histopathological findings or typical imaging features as reference standard.

SECONDARY OUTCOMES:
Comparison of primary and metastatic lesions between [68Ga]Ga-Trivehexin PET/CT and [18F]FDG PET/CT | 2 years
  1. Comparison of tracer uptake values of primary and metastatic lesions between [68Ga]Ga-Trivehexin PET/CT and [18F]FDG PET/CT.
  2. Evaluation of the correlation between [68Ga]Ga-Trivehexin-derived parameters and tumor integrin β6 expression.

CONTACTS AND LOCATIONS:
Overall Officials: Yong He, MD, PhD, Principal Investigator — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kimura RH, Wang L, Shen B, Huo L, Tummers W, Filipp FV, Guo HH, Haywood T, Abou-Elkacem L, Baratto L, Habte F, Devulapally R, Witney TH, Cheng Y, Tikole S, Chakraborti S, Nix J, Bonagura CA, Hatami N, Mooney JJ, Desai T, Turner S, Gaster RS, Otte A, Visser BC, Poultsides GA, Norton J, Park W, Stolowitz M, Lau K, Yang E, Natarajan A, Ilovich O, Srinivas S, Srinivasan A, Paulmurugan R, Willmann J, Chin FT, Cheng Z, Iagaru A, Li F, Gambhir SS. Evaluation of integrin alphavbeta6 cystine knot PET tracers to detect cancer and idiopathic pulmonary fibrosis. Nat Commun. 2019 Oct 14;10(1):4673. doi: 10.1038/s41467-019-11863-w. PMID 31611594
- [Background] Roesch S, Lindner T, Sauter M, Loktev A, Flechsig P, Muller M, Mier W, Warta R, Dyckhoff G, Herold-Mende C, Haberkorn U, Altmann A. Comparison of the RGD Motif-Containing alphavbeta6 Integrin-Binding Peptides SFLAP3 and SFITGv6 for Diagnostic Application in HNSCC. J Nucl Med. 2018 Nov;59(11):1679-1685. doi: 10.2967/jnumed.118.210013. Epub 2018 Apr 19. PMID 29674419
- [Background] Flechsig P, Lindner T, Loktev A, Roesch S, Mier W, Sauter M, Meister M, Herold-Mende C, Haberkorn U, Altmann A. PET/CT Imaging of NSCLC with a alphavbeta6 Integrin-Targeting Peptide. Mol Imaging Biol. 2019 Oct;21(5):973-983. doi: 10.1007/s11307-018-1296-6. PMID 30671741
- [Background] Hausner SH, Bold RJ, Cheuy LY, Chew HK, Daly ME, Davis RA, Foster CC, Kim EJ, Sutcliffe JL. Preclinical Development and First-in-Human Imaging of the Integrin alphavbeta6 with [18F]alphavbeta6-Binding Peptide in Metastatic Carcinoma. Clin Cancer Res. 2019 Feb 15;25(4):1206-1215. doi: 10.1158/1078-0432.CCR-18-2665. Epub 2018 Nov 6. PMID 30401687
- [Background] Keat N, Kenny J, Chen K, Onega M, Garman N, Slack RJ, Parker CA, Lumbers RT, Hallett W, Saleem A, Passchier J, Lukey PT. A Microdose PET Study of the Safety, Immunogenicity, Biodistribution, and Radiation Dosimetry of 18F-FB-A20FMDV2 for Imaging the Integrin alphavbeta6. J Nucl Med Technol. 2018 Jun;46(2):136-143. doi: 10.2967/jnmt.117.203547. Epub 2018 Feb 2. PMID 29438002
- [Background] Van Aarsen LA, Leone DR, Ho S, Dolinski BM, McCoon PE, LePage DJ, Kelly R, Heaney G, Rayhorn P, Reid C, Simon KJ, Horan GS, Tao N, Gardner HA, Skelly MM, Gown AM, Thomas GJ, Weinreb PH, Fawell SE, Violette SM. Antibody-mediated blockade of integrin alpha v beta 6 inhibits tumor progression in vivo by a transforming growth factor-beta-regulated mechanism. Cancer Res. 2008 Jan 15;68(2):561-70. doi: 10.1158/0008-5472.CAN-07-2307. PMID 18199553
- [Background] Elayadi AN, Samli KN, Prudkin L, Liu YH, Bian A, Xie XJ, Wistuba II, Roth JA, McGuire MJ, Brown KC. A peptide selected by biopanning identifies the integrin alphavbeta6 as a prognostic biomarker for nonsmall cell lung cancer. Cancer Res. 2007 Jun 15;67(12):5889-95. doi: 10.1158/0008-5472.CAN-07-0245. PMID 17575158
- [Background] Debordeaux F, Chansel-Debordeaux L, Pinaquy JB, Fernandez P, Schulz J. What about alphavbeta3 integrins in molecular imaging in oncology? Nucl Med Biol. 2018 Jul-Aug;62-63:31-46. doi: 10.1016/j.nucmedbio.2018.04.006. Epub 2018 May 4. PMID 29807242
- [Background] Brzozowska E, Deshmukh S. Integrin Alpha v Beta 6 (alphavbeta6) and Its Implications in Cancer Treatment. Int J Mol Sci. 2022 Oct 15;23(20):12346. doi: 10.3390/ijms232012346. PMID 36293202
- [Background] Quigley NG, Steiger K, Hoberuck S, Czech N, Zierke MA, Kossatz S, Pretze M, Richter F, Weichert W, Pox C, Kotzerke J, Notni J. PET/CT imaging of head-and-neck and pancreatic cancer in humans by targeting the "Cancer Integrin" alphavbeta6 with Ga-68-Trivehexin. Eur J Nucl Med Mol Imaging. 2022 Mar;49(4):1136-1147. doi: 10.1007/s00259-021-05559-x. Epub 2021 Sep 24. PMID 34559266
- [Derived] Wang B, Jiang Y, Zhu J, Wu H, Wu J, Li L, Huang J, Xiao Z, He Y. Fully-automated production of [68Ga]Ga-Trivehexin for clinical application and its biodistribution in healthy volunteers. Front Oncol. 2024 Aug 2;14:1445415. doi: 10.3389/fonc.2024.1445415. eCollection 2024. PMID 39156699